CLINICAL TRIAL: NCT03138395
Title: Predicting Disease Relapse by Monitoring Circulating Cancer DNA After Chemotherapy in Patients With MDS and AML
Brief Title: iCare3: Monitoring Circulating Cancer DNA After Chemotherapy in MDS and AML
Acronym: iCare3
Status: Withdrawn | Type: Observational
Why Stopped: Study design modified to collect specimens from a bank requiring a separate IRB-approved protocol.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201700351; iCare3 (Other: University of Florida); 15963 (Other: University of Florida)
Record Dates: First submitted 2017-04-25; First posted 2017-05-03 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Acute Leukemia; Myelodysplastic Syndromes; AML; MDS
Keywords: acute myeloid leukemia; myelodysplastic syndrome; relapse; PCR; droplet digital; polymerase chain reaction
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * venipuncture peripheral blood
  * bone marrow
  * finger stick peripheral blood
  * saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Specimen Collection: Collection of peripheral blood and bone marrow samples will occur during routine care procedures. Collection of finger stick and saliva specimens will occur on the same day as the peripheral blood and bone marrow procedure, or during routine clinical procedures.
  Interventions: Diagnostic Test: droplet digital PCR

INTERVENTIONS:
Diagnostic Test: droplet digital PCR — This study will use our droplet digital PCR (ddPCR) method to quantify and track peripheral blood plasma MAF in MDS and AML patients before, during and after chemotherapy treatment. Quantification of MAF from fingersticks and saliva samples will also be performed to determine feasibility of obtaining adequate circulating tumor DNA (ctDNA) for ddPCR. Results from this project will generate a non-invasive means to monitor cancer response and progression months before current clinical methods, and provide an opportunity to intervene before the patient relapses.
  Other Names: ddPCR

SUMMARY:
This study will use droplet digital PCR (ddPCR) method to quantify and track peripheral blood plasma mutant allele frequency (MAF) in MDS and AML patients before, during and after chemotherapy treatment. Quantification of MAF from fingersticks and saliva samples will also be performed to determine feasibility of obtaining adequate circulating tumor DNA (ctDNA) for ddPCR.

DETAILED DESCRIPTION:
The greatest challenge in cancer is relapsed disease. Despite best available therapies, approximately 20% of acute myeloid leukemia (AML) patients and 80% of myelodysplastic syndrome (MDS) patients die of relapsed disease. Minimal residual disease (MRD) is the main predictor of refractory disease following chemotherapy. In AML and MDS patients, mutant allele frequency (MAF) associates with future occurrence of relapse. Current oncology practice relies on painful bone marrow biopsies and light microscopy to monitor disease progression, remission, and relapse. Because of the bias in disease sampling and low sensitivity testing, there is an urgent need for a higher sensitivity test to monitor the tumor burden in these patients. The Investigator developed a rapid and ultrahigh sensitivity method to detect cancer-associated mutant alleles. This study will use our droplet digital PCR (ddPCR) method to quantify and track peripheral blood plasma MAF in MDS and AML patients before, during and after chemotherapy treatment. Quantification of MAF from fingersticks and saliva samples will also be performed to determine feasibility of obtaining adequate circulating tumor DNA (ctDNA) for ddPCR. Results from this project will generate a non-invasive means to monitor cancer response and progression months before current clinical methods, and provide an opportunity to intervene before the patient relapses. Furthermore, establishing a quantitative method to measure cancer burden will empower clinical researchers to measure biological activity in phase II and III clinical trials of new therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MDS or AML;
* Have previously consented or prospectively consent to participate in iCare for Cancer (IRB201500073) and the Malignant Hematology Bank (IRB201501063); and
* Must be 18 years of age or older.

Exclusion Criteria:

* Have not previously consented or prospectively consent to participate in iCare for Cancer (IRB201500073) and the Malignant Hematology Bank (IRB201501063); and
* Must be 100 years of age or less.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: AML and MDS patients who have already consented or prospectively consent to participate on iCare for Cancer (IRB 201500073) and the Malignant Hematology Bank (IRB 201501063) to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-09-15 (Estimated); Primary Completion 2018-02-15 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Number of Myeloid Mutations | 1 year
  To count the number of myeloid mutations with the use of a droplet digital PCR (ddPCR) method which will quantify and track peripheral blood plasma, finger stick blood sample, and saliva mutant allele frequency (MAF) in myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML) patients before, during and after chemotherapy treatment.

SECONDARY OUTCOMES:
Number of Myeloid Mutations in circulating DNA tumor (ctDNA) mutations | 1 year
  To count the number myeloid mutations in ctDNA through the collection of serial samples from AML and MDS patients to determine minimal residual disease (MRD) or relapse free survival.
Mutant Allele Frequency (MAF) Ratio | 1 year
  To count the overall number of finger stick and saliva ctDNA MAF and compare it to the overall number of peripheral blood and bone marrow MAF.

CONTACTS AND LOCATIONS:
Overall Officials: Leylah Drusbosky, PhD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No